CLINICAL TRIAL: NCT03922802
Title: Locomotor Function Following Acute Intermittent Hypoxia (AIH) and Transcutaneous Electrical Spinal Cord Stimulation (tSCS) With Gait Therapy Versus Traditional Gait Therapy in Individuals With Spinal Cord Injury
Brief Title: SCI Acute Intermittent Hypoxia and Non-Invasive Spinal Stimulation Combined With Gait Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Director Max Nader Laboratory, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU00211806
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: Spinal Cord Injury; Stimulation; Spinal Stimulation; Noninvasive stimulation; Acute intermittent hypoxia; Hypoxia
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Hypoxia | interventions — Insemination, Artificial, Homologous; Gait

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training (Experimental): May receive up to 45 minutes of AIH prior to up to 50 min of locomotion training with transcutaneous spinal cord stimulation. However, the amount of time spent in side-lying locomotion training, treadmill training and overground training will depend on individual tolerance and progression.
  Intervention: Device: AIH prior to Noninvasive spinal stimulation during gait training
  Interventions: Device: Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training
- Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training (Sham Comparator): May receive up to 45 minutes of Sham AIH prior to up to 50 min of locomotion training with transcutaneous spinal cord stimulation. However, the amount of time spent in side-lying locomotion training, treadmill training and overground training will depend on individual tolerance and progression.
  Interventions: Other: Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training
- Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training (Sham Comparator): May receive up to 45 minutes of Sham AIH prior to up to 50 min of locomotion training with sham transcutaneous spinal cord stimulation. However, the amount of time spent in side-lying locomotion training, treadmill training and overground training will depend on individual tolerance and progression.
  Interventions: Other: Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training

INTERVENTIONS:
Device: Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training — Subjects will receive up to 45 minutes of AIH prior to receiving transcutaneous electrical spinal cord stimulation delivered by a Transcutaneous Spinal Cord Neurostimulator while performing locomotor activities.
  Other Names: AIH + tSCS+ Gait
  Arms: Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training
Other: Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training — Subjects will perform locomotor activities with transcutaneous electrical spinal cord stimulation after receiving sham acute intermittent hypoxia
  Other Names: SHAM AIH + tSCS + Gait
  Arms: Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training
Other: Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training — Subjects will perform locomotor activities with sham transcutaneous electrical spinal cord stimulation after receiving sham acute intermittent hypoxia
  Other Names: SHAM AIH + SHAM tSCS + Gait
  Arms: Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training

SUMMARY:
This is a single blind, sham controlled crossover trial that will evaluate the effectiveness of acute intermittent hypoxia therapy (AIH) combined with transcutaneous (non-invasive) spinal cord stimulation on gait and balance function for individuals after spinal cord injury.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether acute intermittent hypoxia therapy (AIH) combined with transcutaneous spinal cord stimulation during ambulation training modulates spinal locomotor networks in individuals with spinal cord injury
* To determine whether acute intermittent hypoxia therapy (AIH) combined with transcutaneous spinal cord stimulation during ambulation training improves locomotor function in individuals with spinal cord injury
* To determine whether acute intermittent hypoxia therapy (AIH) combined with transcutaneous spinal cord stimulation during ambulation training improves symmetry of gait in individuals with spinal cord injury
* To determine whether acute intermittent hypoxia therapy (AIH) combined with transcutaneous spinal cord stimulation during ambulation training improves standing posture and balance in individuals with spinal cord injury
* To determine whether ambulation efficiency (improved cardiovascular conditioning) improves with a combination of AIH, transcutaneous spinal cord stimulation and ambulation training in individuals with spinal cord injury

ELIGIBILITY:
Inclusion Criteria:

* Participants have been diagnosed with a spinal cord injury below level C2
* ASIA Impairment Scale Grade A-D
* Participants are 18 years of age or older
* Participants are at least 6 months post spinal cord injury
* Participants with paraplegia or tetraplegia secondary to a single spinal cord injury
* Participants are able to provide informed consent
* Participants are not currently receiving regular physical therapy services

Exclusion Criteria:

* Individuals less than 18 years of age
* Individuals less than 6 months post spinal cord injury
* Individuals with ataxia
* Individuals with multiple spinal cord injury history
* Pregnancy or nursing
* Pacemaker or anti-spasticity implantable pumps
* Active pressure sores
* Unhealed bone fractures
* Peripheral neuropathies
* Painful musculoskeletal dysfunction due to active injuries or infections
* Severe contractures in the lower extremities
* Active urinary tract infection
* Clinically significant depression, psychiatric disorders, or ongoing drug abuse
* Diagnosed with any of the following medical conditions: congestive heart failure, cardiac arrhythmias, uncontrolled hypertension, uncontrolled diabetes mellitus, chronic obstructive pulmonary disease, emphysema, severe asthma, previous myocardial infraction, or known carotid/intracerebral artery stenosis
* Individuals with a tracheostomy or who utilize mechanical ventilation.
* Individuals who are currently enrolled in another interventional research study or in therapy related to upper extremity function.
* Participants will be excluded if they have had a botulinum toxin injection to lower extremity musculature within the last 3 months. Participants will need to refrain from lower extremity botulinum toxin injections for the duration of the study. If participants wean off antispasticity medications to successfully complete the responsiveness to AIH screening session, they will need to refrain from the medications for the duration of the study.
* Documented sleep apnea.
* Orthopedic injuries or surgeries that would impact an individual's ability to use the lower extremity.
* Traumatic brain injury or other neurological conditions that would impact the study.
* Blood hemoglobin levels less than 10g/dL.

We will not include the following populations:

* Adults unable to consent, unless accompanied by a legally authorized representative.
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants completed all arms of the study. The order of arm completion was randomly assigned using a block style approach.
Groups:
- All Study Participants: All participants completed 3 arms of the study, in a random order: 1) Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training, 2) Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training, 3) Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training
Period: Overall Study
Arm/Group | All Study Participants
Started | 14
Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | 10
Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | 10
Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training | 10
Completed | 10
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: 10 participants completed and analyzed. 1 was dropped from analysis as an outlier (difference of greater than 1.5*IQR (interquartile range) for all gait outcomes) = 9 participants in analysis total.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.90 (16.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Gait Speed as measured by the 10-meter walk test (10MWT) at self-selected velocity (SSV [Mean (Standard Deviation); unit: meters per second (m/s)] | 0.63 (0.30)

OUTCOME MEASURES:

1. Primary Outcome: Change in 6 Minute Walk Test
Description: The 6 Minute Walk Test (6MWT) measures the distance a subject can walk indoors on a flat, hard surface in a period of 6 minutes, using assertive devices, as necessary. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. This test was completed at 4 time points within each arm: 1) Baseline prior to starting each arm, 2) intervention session 5 within each arm (T5), 3) 3 days after the intervention sessions were complete for the given arm (POST), and 4) 1 week after all intervention sessions were complete for a given arm (1-week follow up)
Time Frame: Baseline (initial visit within an arm), Intervention session 5 within each arm (T5), 3 days after intervention sessions complete within each arm (POST), 1 week after intervention sessions are complete within each arm (1-week follow up)
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: meters (m)
Groups:
- Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training: May receive up to 45 minutes of AIH prior to up to 50 min of locomotion training with transcutaneous spinal cord stimulation. However, the amount of time spent in side-lying locomotion training, treadmill training and overground training will depend on individual tolerance and progression.
  Intervention: Device: AIH prior to Noninvasive spinal stimulation during gait training
  Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training: Subjects will receive up to 45 minutes of AIH prior to receiving transcutaneous electrical spinal cord stimulation delivered by a Transcutaneous Spinal Cord Neurostimulator while performing locomotor activities.
Arm/Group | Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training
Number analyzed (Participants) | 9 | 9 | 9
meters (m)
  Baseline to T5 (7-8 days after baseline from stated arm) | 19.57 [3.68 to 35.46] | 12.28 [-1.58 to 26.13] | 9.63 [-6.45 to 25.71]
  Baseline to POST (10-11 days after baseline from stated arm) | 19.03 [2.94 to 35.13] | 12.01 [-7.41 to 31.44] | 15.63 [6.29 to 24.98]
  Baseline to 1-week follow up (17-19 days after baseline from stated arm) | 21.80 [3.50 to 40.10] | 10.33 [-8.33 to 29.00] | 16.13 [-0.36 to 32.62]

2. Secondary Outcome: Change in 10 Meter Walk Test, Fast Velocity
Description: This test will examine the patient's gait speed. Patients will be directed to walk at their preferred maximum but safe speed: 1) Baseline prior to starting each arm, 2) intervention session 5 within each arm (T5), 3) 3 days after the intervention sessions were complete for the given arm (POST), and 4) 1 week after all intervention sessions were complete for a given arm (1-week follow up)
Time Frame: as for outcome 1
Population: 14 participants enrolled. 4 dropped out of the study due to personal or transportation reasons; therefore, 10 participants completed and analyzed. 1 was dropped from analysis as an outlier (difference of greater than 1.5*IQR (interquartile range) for all gait outcomes) = 9 participants in analysis total.
Measure: Mean (95% Confidence Interval); unit: meters per second
Arm/Group | Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training
Number analyzed (Participants) | 9 | 9 | 9
meters per second
  Baseline to T5 (7-8 days after baseline from stated arm) | 0.03 [-0.02 to 0.08] | 0.00 [-0.05 to 0.04] | 0.04 [-0.01 to 0.10]
  Baseline to POST (10-11 days after baseline from stated arm) | 0.05 [0.01 to 0.09] | -0.01 [-0.07 to 0.05] | 0.02 [-0.02 to 0.07]
  Baseline to 1-week follow up (17-19 days after baseline from stated arm) | 0.03 [-0.03 to 0.10] | 0.01 [-0.09 to 0.12] | -0.01 [-0.08 to 0.05]

3. Secondary Outcome: Timed Up and Go Test: Assesses Mobility, Balance, Walking Ability and Fall Risk
Description: The participant starts seated in a chair with his/her back against the chair back. On command, the participant rises from the chair, walks 3 meters, turns, walks back to the chair and sits down. Timing begins when the command to start is given and stops when the participant returns to a seated position. 1) Baseline prior to starting each arm, 2) intervention session 5 within each arm (T5), 3) 3 days after the intervention sessions were complete for the given arm (POST), and 4) 1 week after all intervention sessions were complete for a given arm (1-week follow up)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training
Number analyzed (Participants) | 9 | 9 | 9
seconds
  Baseline to T5 (7-8 days after baseline from stated arm) | 2.67 [0.18 to 5.16] | 1.45 [-0.94 to 3.84] | 1.00 [0.00 to 2.00]
  Baseline to POST (10-11 days after baseline from stated arm) | 3.39 [1.10 to 5.68] | -0.06 [-1.42 to 1.31] | 0.73 [-0.75 to 2.20]
  Baseline to 1-week follow up (17-19 days after baseline from stated arm) | 3.49 [0.56 to 6.43] | 0.78 [-0.51 to 2.06] | 0.19 [-1.50 to 1.88]

ADVERSE EVENTS:
Time Frame: Baseline to 1-week follow up of third intervention arm (4 months)
Description: Adverse events and serious adverse events were defined as described in the clinicaltrials.gov definitions
Arm/Group | Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | Sham Acute Intermittent Hypoxia + Non Invasive Spinal Cord Stimulation + Gait Training | Sham Acute Intermittent Hypoxia + Sham Non Invasive Spinal Cord Stimulation + Gait Training
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT03922802/Prot_SAP_002.pdf